CLINICAL TRIAL: NCT03331549
Title: Study the High-sensitivity Troponin 0h/1h for Rapid Diagnosis of Non-ST-segment Elevation Myocardial Infarction in the Chinese Population
Brief Title: Study on High-sensitivity Troponin 0h/1h for Rapid Diagnosis of Non-ST-segment Elevation Myocardial Infarction in the Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beckman Coulter, Inc. (Industry)
Responsible Party: Principal Investigator, Shao-Ping Nie, Director, Emergency & Critical Care Center, Professor of Medicine, Beijing Anzhen Hospital
Other Study IDs: 2017020
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Non-ST-segment Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myocardial infarction
- Control group

SUMMARY:
The purpose of the study is to establish a high-sensitivity troponin 0h/1h process for the diagnosis of patients suspected of NSTEMI for the Chinese population, obtain the inclusion and exclusion criteria for diagnosis of these patients and compare the new process with the existing diagnosing methods and processes, including the 3h and 6h processes more extensively used at present and the ECG combined with troponin diagnosis, so as to explore a confirmation model suitable for the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients experiencing acute chest pain or angina pectoris symptom within 12 hours before visiting the hospital;
2. Or those experiencing acute chest pain or angina pectoris peak within 12 hours before visiting the hospital.

Exclusion Criteria:

Patients showing ST-segment elevation during ECG and pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients visiting the Emergency Department of our hospital and have non-traumatic chest pain or other symptoms suggesting acute myocardial infarction will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of non-ST-segment elevation myocardial infarction | After measuring the high-sensitivity troponin level at 1h or 3h

SECONDARY OUTCOMES:
Cardiovascular events or death | Follow-up for 6 months after diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China